CLINICAL TRIAL: NCT04173143
Title: Effects of Cranio- Cervical Flexion Training With and Without Pressure Biofeedback in Patients With Mechanical Neck Pain
Brief Title: Cranio- Cervical Flexion Training With and Without Pressure Biofeedback in Mechanical Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RiphahIU Rabia Ashfaq
Record Dates: First submitted 2019-11-20; First posted 2019-11-21 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Mechanical Neck Pain
Keywords: endurance training,

STUDY DESIGN:
Intervention Model Description: Both experimental and control groups will be treated simultaneously with different modes of endurance training
Who Masked: Participant
Masking Description: This study will be single blinded randomized control trail, participants will be unaware of treatment groups, they will be randomly allocated through sealed envelope method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): This group will receive Cranio cervical flexion training with pressure biofeedback protocol.
  Interventions: Device: Craniocervical flexion training with pressure biofeedback
- Group 2 (Active Comparator): This group will receive Cranio cervical flexion training without pressure biofeedback protocol
  Interventions: Other: Craniocervical flexion training without pressure biofeedback

INTERVENTIONS:
Device: Craniocervical flexion training with pressure biofeedback — Total 15 patients participated in this training group. Session was performed thrice in a week. Each session was givenfor approximately 20minutesPatients were asked to lie in supine hook lying position. After that Pressure biofeedback unit's air bag was clipped together and folded in three and positioned behind the neck just below the occiput. Patients were advised to perform Craniocervical flexion and practiced head nodding action to progressively target (reach the incremental targets) and hold the 5 pressure levels for 10 second between 22 mm Hg and 30 mmHg. A 2 minute second rest period was provided between each level. Minimum performance requirement was 26 mm Hg while ideal performance targets are 28 and 30 mm Hg... Patient will be re-assessed for all baseline variables after 4 weeks of training
  Arms: Group 1
Other: Craniocervical flexion training without pressure biofeedback — Total 15 patients participated in this control group.Session was given 3 times in a week. Each session continue forapproximately 20 minutes. The patient lies in supine crook lying position. The patientwas maximally retracted the chin and asked to maintained it while the patient lifts the head and neck until the head is relatively 2 to 5 cm (1 inch) abovethe couch. The examiner places a hand under the head of patient on the table. Patients were instructed to perform10 repetitions for a hold of 20 seconds initially, increasing it by 10 seconds progressively.The entire session had a maximum of 4 sets. Patient will be re-assessed for all baseline variables after 4 weeks of training
  Arms: Group 2

SUMMARY:
The superficial neck flexor musculature has been given considerate amount of attention to explore its effects on the cervical pain in several researches.. This study intends to put through the benefits of deep cervical flexor training for treatment of cervical neck pain patients.This study will also compare the effects of Cranio cervical flexion training with and without pressure biofeedback on neck pain, muscular endurance,forward head posture and cervical mobility in mechanical neck pain.

DETAILED DESCRIPTION:
The study is Randomized Control Trail, which is being conducted in physical therapy Outpatient department of Pakistan Railway hospital. Sample size of 24 individual was calculated using Epitool with 95% confidence interval (CI) and power 80%. Individual will be screened out according to inclusion criteria. Individuals will be allocated randomly into two groups, 12 in Craniocervical flexion training with pressure biofeedbackgroup and 12 in Craniocervical flexion training without pressure biofeedbackgroup by sealed envelope method.

Deep neck flexor endurance techniquewas used totrain theCraniocervical flexor muscles in control group.Craniocervical flexion technique with Pressure biofeedback unit's was positioned behind the neck just below the occiput was used to train the endurance of the Craniocervical flexor muscle in experimental group.

Assessment will be done on baseline and 4th week. Data will be analyzed on SPSS version 21.

ELIGIBILITY:
Inclusion Criteria:

* • Patients with Chronic mechanical neck pain for more than 3 months duration

  * subjects with aged 25-40 years
  * Numeric pain rating scale (NRPS) greater than 3.
  * Patients with Forward neck posture and a Craniovertebral angle less than 48°

Exclusion Criteria:

* • History of neck surgery, cervical trauma Spinal cord compression, Spinal tumor, Spinal instability

  * History of Spinal fracture, inflammatory disease of spine, Spinal infections, significant neurological deficit, Congenital or acquired postural deformity, doing prescribed exercise for cervical spine.
  * Neck or shoulder pain from non-musculoskeletal causes, demonstrated neurological signs, or had a history of malignancy, current pregnancy.

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Numeric pain rating scale (NPRS) | Baseline
  Numeric pain rating scale (NPRS) is an 11 point (0-10) Scale used to measure pain. Patient verbally select value between (0-10) on the basis of intensity of pain. (0) means No pain and (10) means maximum pain experienced at baseline.
Numeric pain rating scale (NPRS) | Post 4 week
  Numeric pain rating scale (NPRS) is an 11 point (0-10) Scale used to measure pain. Patient verbally select value between (0-10) on the basis of intensity of pain. (0) means No pain and (10) means maximum pain experienced at baseline.
Numeric pain rating scale (NPRS) | Post 6 week
  Numeric pain rating scale (NPRS) is an 11 point (0-10) Scale used to measure pain. Patient verbally select value between (0-10) on the basis of intensity of pain. (0) means No pain and (10) means maximum pain experienced at baseline.
CROM-Flexion | Baseline
  A cervical range of motion (CROM) goniometer will be used to assess cervical range of motion in flexion, extension. Participants will be seated upright and asked to actively move their neck in each direction.
CROM-Flexion | Post 4 week
  A cervical range of motion (CROM) goniometer will be used to assess cervical range of motion in flexion, extension. Participants will be seated upright and asked to actively move their neck in each direction.
CROM-Flexion | Post 6th Week
  A cervical range of motion (CROM) goniometer will be used to assess cervical range of motion in flexion, extension. Participants will be seated upright and asked to actively move their neck in each direction.
CROM-Extention | Baseline
  A cervical range of motion (CROM) goniometer will be used to assess cervical range of motion in flexion, extension. Participants will be seated upright and asked to actively move their neck in each direction.
CROM-Extention | Post 4th Week
  A cervical range of motion (CROM) goniometer will be used to assess cervical range of motion in flexion, extension. Participants will be seated upright and asked to actively move their neck in each direction.
CROM-Extention | Post 6th Week
  A cervical range of motion (CROM) goniometer will be used to assess cervical range of motion in flexion, extension. Participants will be seated upright and asked to actively move their neck in each direction.
Deep neck Flexor endurance | Baseline
  Deep neck flexor endurance test: (Clinical test of endurance for control group)
Deep neck Flexor endurance | Post 4th Week
  Deep neck flexor endurance test: (Clinical test of endurance for control group)
Deep neck Flexor endurance | Post 6th Week
  Deep neck flexor endurance test: (Clinical test of endurance for control group)
Craniocervical flexion test (Clinical test of endurance for experimental group) | Baseline
  The cranio cervical flexion test (CCFT) is used to assess endurance of the deep cervical flexors. A pressure biofeedback unit is inflated to 20 mmHg and is placed behind the neck. While keeping the back of the head stable, the patient performs cranial cervical flexion in a graded fashion in 5 increments (22, 24, 26, 28, and 30 mmHg). Each position is held for 10 seconds with 10 seconds rest between increments.. The test is ended when the pressure decreases >20% or when substitution occurs during the head nod.
Craniocervical flexion test (Clinical test of endurance for experimental group) | Post 4th week
  The cranio cervical flexion test (CCFT) is used to assess endurance of the deep cervical flexors. A pressure biofeedback unit is inflated to 20 mmHg and is placed behind the neck. While keeping the back of the head stable, the patient performs cranial cervical flexion in a graded fashion in 5 increments (22, 24, 26, 28, and 30 mmHg). Each position is held for 10 seconds with 10 seconds rest between increments.. The test is ended when the pressure decreases >20% or when substitution occurs during the head nod.
Craniocervical flexion test (Clinical test of endurance for experimental group) | Post 6th week
  The cranio cervical flexion test (CCFT) is used to assess endurance of the deep cervical flexors. A pressure biofeedback unit is inflated to 20 mmHg and is placed behind the neck. While keeping the back of the head stable, the patient performs cranial cervical flexion in a graded fashion in 5 increments (22, 24, 26, 28, and 30 mmHg). Each position is held for 10 seconds with 10 seconds rest between increments.. The test is ended when the pressure decreases >20% or when substitution occurs during the head nod.

SECONDARY OUTCOMES:
Cranio-vertebral angle | Baseline
  On protractor tool was used to measure forward head posture through a craniovertebral angle (CVA).. It has excellent reliability value (ICC 0.991).Participants were asked to sit on a stool and concentrate at a specific point on their eye level.Then we used three markers: one on C7, the other on tragus and the third on canthus. The angle between the line connecting C7 to tragus and a vertical line extending from C7 was calculated and images were taken. Patients having a Craniovertebral angle less than 48°were considered in category of forward head posture.
Cranio-vertebral angle | Post 4th week
  On protractor tool was used to measure forward head posture through a craniovertebral angle (CVA).. It has excellent reliability value (ICC 0.991).Participants were asked to sit on a stool and concentrate at a specific point on their eye level.Then we used three markers: one on C7, the other on tragus and the third on canthus. The angle between the line connecting C7 to tragus and a vertical line extending from C7 was calculated and images were taken. Patients having a Craniovertebral angle less than 48°were considered in category of forward head posture.
Cranio-vertebral angle | Post 6th week
  On protractor tool was used to measure forward head posture through a craniovertebral angle (CVA).. It has excellent reliability value (ICC 0.991).Participants were asked to sit on a stool and concentrate at a specific point on their eye level.Then we used three markers: one on C7, the other on tragus and the third on canthus. The angle between the line connecting C7 to tragus and a vertical line extending from C7 was calculated and images were taken. Patients having a Craniovertebral angle less than 48°were considered in category of forward head posture.

CONTACTS AND LOCATIONS:
Overall Officials: Huma Riaz, PHD*, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Railway hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gupta BD, Aggarwal S, Gupta B, Gupta M, Gupta N. Effect of Deep Cervical Flexor Training vs. Conventional Isometric Training on Forward Head Posture, Pain, Neck Disability Index In Dentists Suffering from Chronic Neck Pain. J Clin Diagn Res. 2013 Oct;7(10):2261-4. doi: 10.7860/JCDR/2013/6072.3487. Epub 2013 Oct 5. PMID 24298492
- [Background] Kim JY, Kwag KI. Clinical effects of deep cervical flexor muscle activation in patients with chronic neck pain. J Phys Ther Sci. 2016 Jan;28(1):269-73. doi: 10.1589/jpts.28.269. Epub 2016 Jan 30. PMID 26957772
- [Background] Kang DY. Deep cervical flexor training with a pressure biofeedback unit is an effective method for maintaining neck mobility and muscular endurance in college students with forward head posture. J Phys Ther Sci. 2015 Oct;27(10):3207-10. doi: 10.1589/jpts.27.3207. Epub 2015 Oct 30. PMID 26644676
- [Background] Iqbal ZA, Rajan R, Khan SA, Alghadir AH. Effect of deep cervical flexor muscles training using pressure biofeedback on pain and disability of school teachers with neck pain. J Phys Ther Sci. 2013 Jun;25(6):657-61. doi: 10.1589/jpts.25.657. Epub 2013 Jul 23. PMID 24259822
- [Background] Suvarnnato T, Puntumetakul R, Uthaikhup S, Boucaut R. Effect of specific deep cervical muscle exercises on functional disability, pain intensity, craniovertebral angle, and neck-muscle strength in chronic mechanical neck pain: a randomized controlled trial. J Pain Res. 2019 Mar 7;12:915-925. doi: 10.2147/JPR.S190125. eCollection 2019. PMID 30881101